CLINICAL TRIAL: NCT07319130
Title: Clinical Study of 68Ga-labeled Novel Nectin-4 Bicyclic Peptide PET/CT for Imaging of Solid Tumors With High Nectin-4 Expression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-68Ga-Nectin-4-peptide 02
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors With High Expression of Nectin4
MeSH Terms: interventions — Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Nectin4 bicyclic peptide PET/CT imaging (Experimental)
  Interventions: Diagnostic Test: Immunohistochemistry

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry — Nectin4 Immunohistochemistry testing

SUMMARY:
Tumors are one of the major diseases threatening human health, among which solid tumors account for a considerable proportion. Nectin-4, as an important cell adhesion molecule, shows a highly expressed state in various solid tumors. In triple-negative breast cancer, the high expression rate of Nectin-4 can reach more than 50%, and it is closely associated with tumor invasion, metastasis and poor prognosis. Relevant studies have shown that the five-year survival rate of triple-negative breast cancer patients with high expression of Nectin-4 is significantly lower than that of patients with low expression. In urothelial carcinoma, the positive expression rate of Nectin-4 is also relatively high, reaching 40%-60%, and it is a highly potential target for tumor treatment and diagnosis. Its abnormal expression in solid tumors has opened up a new direction for the early diagnosis and targeted therapy of tumors. However, at present, the precise diagnosis and effective treatment of solid tumors with high expression of Nectin-4 still face many challenges. There is an urgent need for new technologies and methods to improve the diagnosis and treatment level in order to improve the prognosis of patients. Therefore, this study aims to develop a method targeting the Nectin4 bicyclic peptide to achieve non-invasive visualization of Nectin4 expression in tumors. This approach may also contribute to the formulation and optimization of clinical treatment strategies

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 75 years old (including the boundary value), gender not limited. 2. Solid tumors (such as urothelial carcinoma, breast cancer, lung cancer, etc.) that have been pathologically diagnosed with high expression of Nectin-4 within one month before imaging.

  3. At least one evaluable tumor lesion (primary or metastatic) exists. 4. Voluntarily sign the informed consent form and be able to cooperate with the research process.

  5.ECOG score: 0 to 2 points, expected survival period: ≥6 months.

Exclusion Criteria:

* 1. Combined with other active malignant tumors (excluding non-melanoma skin cancer or carcinoma in situ).

  2. Severe heart, liver and kidney insufficiency (such as ALT/AST >3 times ULN, creatinine clearance rate <30 mL/min).

  3. Uncontrolled systemic infections or immune system diseases. 4. Pregnant or lactating women, or patients of childbearing age who have not taken effective contraceptive measures.

  5. Previously received Nectin-4 targeted therapy (such as Enfortumab vedotin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PET/CT imaging SuV value | 0-45 minutes, 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China